CLINICAL TRIAL: NCT03075774
Title: FibCard Study: Observational Study About the Use of Fibrinogen in Adult Cardiac Surgery
Brief Title: Observational Study About the Use of Fibrinogen in Adult Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Collaborators: Keyrus Biopharma (Other)
Responsible Party: Sponsor
Other Study IDs: FibCard-N°RCB : 2016-A01995-46
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Cardiac Surgery; Extracorporeal Circulation; Fibrinogen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter prospective observational study, involving all adult patients who underwent cardiac surgery with extracorporeal circulation

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18 that underwent a cardiac surgery with extracorporeal circulation.
* Patient who agreed to participate in the study.

Exclusion Criteria:

* Patient under the age of 18.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient that underwent a cardiac surgery with extracorporeal circulation.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
The international recommendations published by ESA in 2016 | 13 Months
  Review the concordance between the presence / absence of indication (according to the international recommendations published by ESA in 2016) and the prescription / non-prescription of fibrinogen concentrates

REFERENCES:
- [Derived] Longrois D, Albaladejo P, Bedague D, Ouattara A, Bougle A, Dureau P, Cholley B, Mertes PM, Provenchere S, Robin E, Besch G, Grelet T, Grosjean S, Guinot PG, Rozec B, Rigal JC, Fellahi JL, Colson P; SFAR Research Committee. Compliance with ESAIC guidelines for fibrinogen concentrate prescription in cardiac surgery: a multicentre French cohort study. BMC Anesthesiol. 2025 Nov 24;25(1):594. doi: 10.1186/s12871-025-03347-w. PMID 41286643